CLINICAL TRIAL: NCT02737384
Title: Hematopoietic Stem Cells Transplantation in Children With Combined Immunodeficiency (CID): Selective Depletion of Naive Cells From the Graft
Brief Title: Hematopoietic Stem Cells Transplantation in Children With Combined Immunodeficiency (CID)
Acronym: CD45RA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P140317; 2015-A01256-43 (Other: ANSM)
Record Dates: First submitted 2016-04-08; First posted 2016-04-13 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-04

CONDITIONS: Combined Immunodeficiencies
Keywords: Combined immunodeficiencies; hematopoietic stem cell transplantation; CD45RA; primitive immunodeficiencies; pediatric transplantation; CD45RA depletion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Biological: Depletion in CD45RA graft donor

INTERVENTIONS:
Biological: Depletion in CD45RA graft donor — Experimental treatment: negative fraction after CD34+ selection from PBSC graft is depleted of naïve CD45RA+ cells. this fraction is reinjected to the recipient and is the experimental product.
  Conditioning regimen:
  Up-front ATG from D-14 toD-11 Busulphan IV from D-8 to -5 Fludarabine from D-7 to D-4 Thiothepa D-3 to D-2
  Graft: CD34+ cells positively selected cells from PBSC of the donor
  Post transplant immunosuppression: ciclosporin started at D-1 to D+100

SUMMARY:
The purpose of this study is to evaluate selective depletion of naïve CD45RA+ T cells from allogenic peripheral blood stem cell graft in children transplanted for combined immune deficiency. The aims of this procedure are to prevent graft versus host disease (GVHD) while preserving anti-infectious response from donor memory T lymphocytes.

DETAILED DESCRIPTION:
Combined immunodeficiencies (CIDs) are an heterogeneous group of primitive immunodeficiency (PID), which affect T cells development, function or both. These inherited conditions can only be cured by allogeneic hematopoietic stem cell transplantation (HSCT). These procedures have a high risk of morbidity and mortality such a graft versus host disease (GVHD), rejection of the graft and serious infections, especially in this population of children with PID. GVHD is more frequent and severe if the donor is not an identical sibling and/or presents an HLA-mismatch. GVHD requires high immunosuppression as prevention and treatment, and therefore impedes immunity against infections.

In vitro and animal models suggest that GVHD is mediated by naïve T cells. The aim of this study is to decrease the rate and severity of GVHD after selective depletion of naïve CD45RA+ T cells from allogeneic hematopoietic stem cell grafts in patients with CIDs with high risk of severe GVHD, and to preserve immunity against pathogens in a population with high vulnerability to infections.

The project aims is, first, to show improvement of rejection-free and GVH-free survival 12 months post-transplant, and secondly, to show the decrease of viral infection, and assess immune reconstitution kinetic and quality and specific antiviral responses, after a engraftment with naïve cell depleted allograft.

ELIGIBILITY:
Inclusion Criteria:

* Patient from 12 months to 18 years
* Combined immunodeficiencies with known molecular diagnosis or if unknown, corresponding of p-CID study's definition
* Hematopoietic stem cell Transplantation planned with one of the following donors :
* sibling with 1 or 2 HLA antigens mismatch
* parent 10/10 or 9/10 identical
* unrelated donor: 10/10 or 9/10 identical
* Consent form signed by the child's legal guardian
* Patient using effectiveness contraception during this trial
* Affiliated or beneficiary of a health insurance regimen

Exclusion Criteria:

* Wiskott-Aldrich syndrome
* Ongoing pregnancy
* Positive HIV PCR
* Contraindication for hematopoetic stem cell transplantation
* Geno-identical donor in the siblings
* hematopoetic stem cell transplantation antecedent

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Number of death | 12 months after the transplantation
Number of graft rejection | 12 months after the transplantation
Number of graft versus host disease (GVHD) grade III or IV | 12 months after the transplantation

SECONDARY OUTCOMES:
Need of antiviral treatment | 12 months after the transplantation
  to assess viral infection
T Lymphocyte proliferations to phytohemagglutinin (PHA) | 12 months after the transplantation
  to assess immune reconstitution
Proportion of T CD4 and CD8 lymphocytes specific of cytomegalovirus, Epstein Barr virus and adenovirus | 12 months after the transplantation
  to assess specific antiviral response

CONTACTS AND LOCATIONS:
Overall Officials: Marina CAVAZZANA, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Touzot F, Neven B, Dal-Cortivo L, Gabrion A, Moshous D, Cros G, Chomton M, Luby JM, Terniaux B, Magalon J, Picard C, Blanche S, Fischer A, Cavazzana M. CD45RA depletion in HLA-mismatched allogeneic hematopoietic stem cell transplantation for primary combined immunodeficiency: A preliminary study. J Allergy Clin Immunol. 2015 May;135(5):1303-9.e1-3. doi: 10.1016/j.jaci.2014.08.019. Epub 2014 Oct 3. PMID 25282016